CLINICAL TRIAL: NCT04330144
Title: A Study of Hydroxychloroquine as Post Exposure Prophylaxis for SARS-CoV-2(HOPE Trial)
Brief Title: Hydroxychloroquine as Post Exposure Prophylaxis for SARS-CoV-2(HOPE Trial)
Acronym: COVID-19
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Goo Song, Professor, Department of Internal Medicine,, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3-2020-0036
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Contact Person From COVID-19 Confirmed Patient
Keywords: Postexposure prophylaxis; hydroxychloroquine; SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Post-Exposure Prophylaxis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- administration of hydroxychloroquine as PEP (Experimental)
  Interventions: Drug: Hydroxychloroquine as post exposure prophylaxis
- control with no PEP (Active Comparator)
  Interventions: Other: Others(No intervention)

INTERVENTIONS:
Drug: Hydroxychloroquine as post exposure prophylaxis — 1day: Hydroxychloroquine 800mg Qd po 2-5dy: Hydroxychloroquine 400mg Qd po
  Arms: administration of hydroxychloroquine as PEP
Other: Others(No intervention) — No treatment. Close monitoring and quarantine.
  Arms: control with no PEP

SUMMARY:
There is no known definite treatment after exposure to SARS-CoV-2, but the some animal and clinical trials confirmed the efficacy of hydroxychloroquine (HCQ) or chloroquine against SARS-CoV-2. Thus, in this study, we aim to evaluate the efficacy and safety of hydroxychloroquine as post exposure prophylaxis for SARS-CoV-2.

* Primary end point: comparison the rate of COVID-19 between PEP with HCQ and control group.
* Secondary end point: Comparison of the rate of COVID-19 according to the contact level (time, place, degree of wearing personal protective equipment).
* Safety comparison: Safety verification by identifying major side effects in the HCQ group."

ELIGIBILITY:
Inclusion Criteria:

* A contact person from confirmed case of SARS-CoV-2 infection
* Medical staff exposed from confirmed case of SARS-CoV-2 infection in hospitals
* Persons exposed to SARS-CoV-2 in COVID-19 outbreak situation with certain workplaces, religious groups, and military, etc.

  * Subjects of study include both symptomatic and asymptomatic contacts.

Exclusion Criteria:

* Hypersensitivity to Chloroquine or Hydroxychloroquine
* Those who are contraindicated in Hydroxychloroquine administration according to the permission requirements such as pregnant women, nursing mothers, visual disorders, macular disease, and porphyria, etc.
* Human immunodeficiency virus (HIV) infected person
* Patients with autoimmune disease (Systemic lupus erythematosus, Mixed connective tissue disease)
* Patients with autoimmune rheumatoid inflammatory disease (AIIRD; Autoimmune inflammatory rheumatic diseases - Ankylosing spondylitis, Rheumatic arthritis, Psoriatic arthritis)
* Arrhythmia, liver cirrhosis of Child Pugh C, chronic renal failure with eGFR≤30mL / min / 1.73m2
* A person who is positive in the COVID-19 screening PCR test before starting PEP

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
The rate of COVID-19 | PCR test of COVID-19 at 14 days after the contact from confirmed case
  After postexposure prophylaxis, the rate of COVID-19 conversion between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Yong Goo Song, Professor, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea